CLINICAL TRIAL: NCT07216742
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of a Human Menopausal Gonadotropin in the Development of Multiple Follicles, Pregnancy, and Cumulative Live Birth as Part of an Assisted Reproductive Technology (ART) Cycle.
Brief Title: Human Menopausal Gonadotropin Research in Infertility Assessing Cumulative Live Birth With Frozen Embryo Transfer.
Acronym: GRACE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Granata Bio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBHMG-301
Record Dates: First submitted 2025-10-02; First posted 2025-10-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Infertility (IVF Patients)
Keywords: Controlled ovarian stimulation; Gonadotropins; frozen embryo transfer; cumulative live birth rate; hMG
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- hMG (Experimental): Human Menopausal Gonadotropin, daily subcutaneous injection
  Interventions: Drug: hMG subcutaneous injection
- Placebo (Placebo Comparator): Placebo, daily subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hMG subcutaneous injection — daily subcutaneous injection
  Arms: hMG
Drug: Placebo — daily subcutaneous injection
  Arms: Placebo

SUMMARY:
The goal of this multicenter, randomized, placebo-controlled, double-blind clinical trial is toto evaluate the efficacy and safety of a human menopausal gonadotropin (hMG) in the development of multiple follicles, pregnancy, and cumulative live birth as part of an Assisted Reproductive Technology (ART) cycle in in women with a diagnosis of infertility.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 18-42 years old at the time of consent.
* BMI ≥18 and <38 kg/m² at the time of consent.
* Menstrual cycles between 21-35 days.
* Normal mammogram or breast ultrasound if patient is >40 or if participant is younger as indicated by physician recommendation, within 2 years of screening.
* Anti-Müllerian hormone (AMH) >1.2 ng/ml within 6 months of screening.
* If donor sperm is used, donor must be 18-40 years of age at the time of collection and compliant with 21 Code of Regulations (CFR) section 1271 Subpart C.
* Transvaginal ultrasound (TVUS) documenting presence and adequate visualization of both ovaries without ovarian enlargement, normal adnexa, and both ovaries accessible for oocyte retrieval at screening or within 6 months of screening.
* Valid medical indication for in vitro fertilization (IVF) treatment and subsequent embryo transfer (i.e. history of infertility according to current American Society of Reproductive Medicine (ASRM) definition, single women or same-sex couples) with the intention to achieve pregnancy within 12 months of the first stimulation cycle.
* Hysterosalpingography, hysteroscopy or saline infusion sonography, documenting a normal uterine cavity (i.e. no müllerian duct anomaly, uterine fibroids, endometrial polyps, intrauterine adhesions, adenomyosis) at screening or within 1 year prior to screening.
* Normal cervical cytology/high risk human papillomavirus (HPV) testing per American College of Obstetrician/Obstetrician Gynecologist (OB/GYN) (ACOG) guidelines.
* Negative serum hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus (HIV) antibody tests at screening.
* Absence of hydrosalpinx confirmed by hysterosalpingogram (HSG), sonohysterogram, laparoscopy, or other appropriate imaging within the past 12 months.
* Willing to undergo up to two ovarian stimulation cycles prior to frozen embryo transfer.
* Willing to self-administer study medications.
* Willing to have trophectoderm biopsy of all blastocyst stage embryos.
* Willing to accept transfer of one euploid embryo.
* Willing to vitrify and warm embryo(s) with intention to have a Frozen Embryo Transfer (FET).
* Willing and able to comply with the protocol and schedule of events for the duration of the study as well as providing delivery data and neonatal health data.

Exclusion Criteria:

* Persistent ovarian cysts (≥11 mm) for >1 cycle or ovarian endometrioma on ultrasound (Principal Investigator's [PI] discretion).
* Participants with hepatic impairment (liver function tests > 2x upper limit of normal). Participants with renal impairment (estimated creatinine clearance <60 mL/min/1.73 m2).
* Uncontrolled adrenal or thyroid dysfunction.
* Greater than one IVF cycle canceled due to inability to meet ovulation trigger criteria (i.e. at least 2-3 follicles reach ≥18 mm.).
* History of recurrent implantation failure (RIF), defined according to the Lugano Consensus as the absence of implantation after transfer of ≥4 good-quality embryos in ≥3 embryo transfer (ET) cycles in women under the age of 40, using autologous oocytes.
* Recurrent pregnancy loss (RPL) is defined by two or more miscarriages; that is clinical pregnancies with the same partner and documented by ultrasonography or histopathological examination.
* Known history of anovulation.
* Antral Follicle Count (AFC) <5 at screening.
* One or more follicles ≥11 mm observed on TVUS prior to randomization on stimulation day 1.
* Past or current history of an estrogen dependent malignancy
* Untreated atypical endometrial hyperplasia
* Any contraindication to the use of oral contraceptives
* History of OHSS.
* Morphological sperm evidence of globozoospermia or prior failed oocyte fertilization in previous IVF cycle.
* The use of donor sperm back up or rescue for fertilization of oocytes.
* Use of calcium ionophore or treatment of sperm with methyl xanthines.
* The need for surgically retrieved sperm (i.e. testicular sperm extraction [TESE], Percutaneous Epididymal Sperm Aspiration [PESA]).
* Use of any investigational drug throughout the study, or within 3 months before screening or 5 half-lives whichever is longer.
* Any concomitant medication that would interfere with the evaluation of the study medication (anti-psychotics, anxiolytics, hypnotics, sedatives, non-study hormonal therapy, except thyroid medication,).
* Current use or dependence on psychotropic medications that are contraindicated during pregnancy or have known or suspected fetal risk
* Required chronic use of non-steroidal anti-inflammatory drugs during cycle.
* Treatment with clomiphene citrate, metformin, gonadotropins, or GnRH analogs within 1 month prior to randomization.
* Pregnancy, lactation, or contraindication to gonadotropins.
* Known thrombophilia or history of blood clots unless fully evaluated and cleared by a hematologist and receiving appropriate prophylaxis.
* Known abnormal karyotype in the patient or her partner that is considered clinically significant, such as numerical or structural chromosomal abnormalities (e.g., translocations, inversions, aneuploidies) known to impair fertility, increase risk of miscarriage, or result in genetic disorders in offspring.
* Current tobacco user.
* Current or past (last 12 months) abuse of alcohol or drugs.
* Current use of dietary supplements containing high dose of biotin (>300µg), if prior use washout period of 1 week prior to randomization.
* No use of bioidentical hormones during stimulation or up to three months prior to start of stimulation. If prior use: washout period of three months prior to being randomized.
* A history of chemotherapy or radiotherapy.
* Undiagnosed uterine bleeding.
* Tumors of the ovary, breast, adrenal gland, pituitary, or hypothalamus; malformation of sexual organs incompatible with pregnancy.
* Known active pelvic inflammatory disease.
* Current, untreated submucosal fibroids or Intramural fibroids ≥5 cm or otherwise clinically relevant pathology that could impair embryo implantation or pregnancy continuation.
* The presence of severe endometriosis (ASRM stage 3 or stage 4) confirmed by laparoscopy, Magnetic Resonance Imaging (MRI), or pelvic ultrasound.
* Concomitant participation in another study protocol.
* Couples identified as carriers of the same autosomal recessive genetic condition associated with serious health outcomes in offspring will be excluded from the trial.
* Planned use of a gestational carrier.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 659 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
cumulative live birth rate | 12 months
  cumulative live birth rate following vitrified-thawed, single-euploid blastocyst transfer(s)

SECONDARY OUTCOMES:
Positive pregnancy (serum β-human chorionic gonadotropin [hCG]) | 10 +/-2 days after Embryo transfer
Clinical pregnancy (intrauterine gestational sac with fetal heartbeat) | 5 weeks ± 6 days post-embryo transfer
Ongoing pregnancy (intrauterine pregnancy with fetal heartbeat) | 10 weeks ± 6 days post-embryo transfer (ET)
Live birth rate | 9 months after ET
Number of oocytes retrieved per stimulation cycle | 12-22 days after controlled ovarian stimulation start
Number of metaphase II (MII) oocytes retrieved | 12-22 days after controlled ovarian stimulation start
Fertilization rate (proportion of MII oocytes with normal fertilization) | 12-22 days after Controlled Ovarian stimulation start
Number of Day 5 blastocysts from oocyte retrievals from Period 1 and Period 2 | 12-22 days after controlled ovarian stimulation start
Total gonadotropin dose required per stimulation cycle | 12-20 days after start Controlled ovarian stimulation
Serum estradiol concentration on the day of ovulation trigger | 12-20 days after controlled ovarian stimulation start
Serum progesterone (P4) on Day 5 of stimulation | 5 days after start controlled ovarian stimulation
Serum Follicular Stimulation Hormone (FSH) level on stimulation day 1, pre-dose | 1 day of stimulation
Serum Luteinizing hormone (LH) level on stimulation day 1, pre-dose | 1 day of stimulation
Serum human Chorionic Gonadotropin (hCG) level on stimulation day 1, pre-dose | 1 day of stimulation
FSH level on stimulation day 1, 1-4 hours post dose | 1 day of stimulation
LH level on stimulation day 1, 1-4 hours post dose | 1 day of stimulation
hCG level on stimulation day 1, 1-4 hours post dose | 1 day of stimulation
FSH level on stimulation day 5 | After 5 day of stimulation
LH level on stimulation day 5 | After 5 day of stimulation
hCG level on stimulation day 5 | After 5 day of stimulation
FSH level on last stimulation day | 12-20 days after controlled ovarian stimulation start
LH level on last stimulation day | 12-20 days after controlled ovarian stimulation start
hCG level on last stimulation day | 12-20 days after controlled ovarian stimulation start
FSH level on oocytes retrieval day | 12-22 days after controlled ovarian stimulation start
LH level on oocytes retrieval day | 12-22 days after controlled ovarian stimulation start
hCG level on oocytes retrieval day | 12-22 days after controlled ovarian stimulation start

OTHER OUTCOMES:
Incidence, severity, timing, and duration of treatment-emergent adverse events (TEAEs), including action taken and outcome | up to 10 weeks post embryo transfer
Injection sites reactions (e.g., pain, erythema, swelling) | 20 days after Controlled ovarian stimulation start
Incidence of early and late ovarian hyperstimulation syndrome (OHSS) | up to 10 weeks post Embryo transfer
Development of treatment-emergent anti-drug antibodies | up to 5 weeks +/- 6 days after embryo transfer
Singleton live birth | 9 months post embryo transfer
Multiple gestations (twins, triplets, or higher-order multifetal pregnancies) | 9 months after Embryo transfer
Biochemical pregnancy loss | up to 6 weeks after embryo transfer
Ectopic pregnancy | Up to 6 weeks after embryo transfer
Early pregnancy loss | Up to 12 weeks of gestation
Intrauterine fetal demise | up to 9 months after embryo transfer
Incidence of maternal/pregnancy complications | up to 9 months after embryo transfer
Preterm birth | up to 37 weeks of gestation
Small for gestational age | up to 9 months after Embryo transfer
Stillbirth | up to 9 months after embryo transfer

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - HRC Fertility, Encino, California
  - Illume Fertility, Norwalk, Connecticut
  - Reproductive Associates of Delaware CCRM, Newark, Delaware
  - IVF Florida Reproductive Associates, Margate, Florida
  - Center for Reproductive Medicine, Winter Park, Florida
  - Reproductive Biology Associates (RBA), Atlanta, Georgia
  - Fertility Institute of Hawaii, Honolulu, Hawaii
  - Fertility Centers of Illinois, Chicago, Illinois
  - Shady Grove Fertility - Rockville, Rockville, Maryland
  - Boston IVF, Waltham, Massachusetts
  - Reach Fertility, Charlotte, North Carolina
  - Carolina Conceptions, Raleigh, North Carolina
  - Pinnacle Fertility - Oregon, Portland, Oregon
  - Main Line Fertility, Bryn Mawr, Pennsylvania
  - CARE Fertility, Bedford, Texas
  - Shady Grove Houston, Webster, Texas

IPD SHARING:
Plan to Share IPD: No